CLINICAL TRIAL: NCT00132782
Title: Relationship Between Functional Health Status and Ventricular Performance After Fontan (A Trial Conducted by the Pediatric Heart Network)
Brief Title: Relationship Between Functional Health Status and Ventricular Performance After Fontan--Pediatric Heart Network
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Lynn Sleeper, ScD., New England Research Institutes
Other Study IDs: 242; U01HL068270 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2009-02

CONDITIONS: Defect, Congenital Heart; Arrhythmia
MeSH Terms: conditions — Heart Defects, Congenital; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this cross-sectional study was to determine the interrelationships between health status and measures of cardiac performance in children 6 to 18 years of age with congenital heart disease who have undergone a Fontan procedure as surgical treatment for functional single ventricle. The goal was to develop a data set that will permit identification of a clinically relevant endpoint for subsequent trials of medical management of the Fontan patient.

DETAILED DESCRIPTION:
BACKGROUND:

Children born with one functional ventricle and who undergo a Fontan procedure, have a higher incidence of late complications than other congenital heart patients. While the Fontan procedure results in restoring near-normal systemic oxygen saturation, there are recognized problems and little information about the overall health status, functional status and ventricular performance in these children.

DESIGN NARRATIVE:

This cross-sectional observational study included children 6-18 years of age who had undergone a Fontan procedure for a congenital cardiac defect. Prospective data collection for each patient occured within a 3 month time period and included cardiac MRI, echocardiography, serology and exercise testing. Historical clinical and surgical data, as well as parent and child self reports of health status, was collected.

ELIGIBILITY:
Inclusion Criteria

* Age 6 through 18 years at the time of enrollment.
* Fontan surgery of any type at least 6 months prior to the time of testing.
* Agreement and ability to have all of the following testing completed:

  1. An echocardiogram at the study center,
  2. Parent health status questionnaire, and
  3. Blood testing.
* Planned or ongoing cardiac care at the study center that will allow completion of study testing within 3 months of study enrollment.
* Informed consent of a parent or guardian, and assent of the study participant if he/she is able to provide it, according to institutional guidelines.

Exclusion Criteria

* Non-cardiac medical or psychiatric disorder that would prevent successful completion of planned study testing or would invalidate the results of study testing.
* Ongoing or planned participation in another research protocol that would either prevent successful completion of planned study testing or invalidate the results of study testing.
* Lack of reading fluency by the primary caregiver in both English and Spanish, languages for which the parental report health status questionnaire has been validated.
* Pregnancy at the time of enrollment or pregnancy planned prior to completion of study testing.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects must have had Fontan surgery of any type at least 6 months prior to the time of testing
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2003-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sleeper, ScD, Principal Investigator — Carelon Research

REFERENCES:
- [Derived] Atz AM, Zak V, Mahony L, Uzark K, D'agincourt N, Goldberg DJ, Williams RV, Breitbart RE, Colan SD, Burns KM, Margossian R, Henderson HT, Korsin R, Marino BS, Daniels K, McCrindle BW; Pediatric Heart Network Investigators. Longitudinal Outcomes of Patients With Single Ventricle After the Fontan Procedure. J Am Coll Cardiol. 2017 Jun 6;69(22):2735-2744. doi: 10.1016/j.jacc.2017.03.582. PMID 28571639
- [Derived] Margossian R, Sleeper LA, Pearson GD, Barker PC, Mertens L, Quartermain MD, Su JT, Shirali G, Chen S, Colan SD; Pediatric Heart Network Investigators. Assessment of Diastolic Function in Single-Ventricle Patients After the Fontan Procedure. J Am Soc Echocardiogr. 2016 Nov;29(11):1066-1073. doi: 10.1016/j.echo.2016.07.016. Epub 2016 Sep 10. PMID 27624592
- [Derived] Uzark K, Zak V, Shrader P, McCrindle BW, Radojewski E, Varni JW, Daniels K, Handisides J, Hill KD, Lambert LM, Margossian R, Pemberton VL, Lai WW, Atz AM; Pediatric Heart Network Investigators. Assessment of Quality of Life in Young Patients with Single Ventricle after the Fontan Operation. J Pediatr. 2016 Mar;170:166-72.e1. doi: 10.1016/j.jpeds.2015.11.016. Epub 2015 Dec 10. PMID 26685073
- [Derived] Atz AM, Zak V, Mahony L, Uzark K, Shrader P, Gallagher D, Paridon SM, Williams RV, Breitbart RE, Colan SD, Kaltman JR, Margossian R, Pasquali SK, Allen K, Lai WW, Korsin R, Marino BS, Mirarchi N, McCrindle BW; Pediatric Heart Network Investigators. Survival data and predictors of functional outcome an average of 15 years after the Fontan procedure: the pediatric heart network Fontan cohort. Congenit Heart Dis. 2015 Jan-Feb;10(1):E30-42. doi: 10.1111/chd.12193. Epub 2014 Jun 17. PMID 24934522
- [Derived] Atz AM, Travison TG, McCrindle BW, Mahony L, Glatz AC, Kaza AK, Breitbart RE, Colan SD, Kaltman JR, Margossian R, Pasquali SK, Wang Y, Gersony WM; Pediatric Heart Network Investigators. Cardiac performance and quality of life in patients who have undergone the Fontan procedure with and without prior superior cavopulmonary connection. Cardiol Young. 2013 Jun;23(3):335-43. doi: 10.1017/S1047951112001175. Epub 2012 Jul 24. PMID 22824161
- [Derived] Cohen MS, Zak V, Atz AM, Printz BF, Pinto N, Lambert L, Pemberton V, Li JS, Margossian R, Dunbar-Masterson C, McCrindle BW. Anthropometric measures after Fontan procedure: implications for suboptimal functional outcome. Am Heart J. 2010 Dec;160(6):1092-8, 1098.e1. doi: 10.1016/j.ahj.2010.07.039. PMID 21146663
- [Derived] Stephenson EA, Lu M, Berul CI, Etheridge SP, Idriss SF, Margossian R, Reed JH, Prakash A, Sleeper LA, Vetter VL, Blaufox AD; Pediatric Heart Network Investigators. Arrhythmias in a contemporary fontan cohort: prevalence and clinical associations in a multicenter cross-sectional study. J Am Coll Cardiol. 2010 Sep 7;56(11):890-6. doi: 10.1016/j.jacc.2010.03.079. PMID 20813285